CLINICAL TRIAL: NCT00700739
Title: A Multi-Centre, Prospective, Randomized, Post Marketing Surveillance Study Comparing Cervical Arthroplasty to Anterior Cervical Discectomy and Fusion (ACDF) for the Treatment of Cervical Degenerative Disc Disease
Brief Title: Study to Investigate the Performance of Cervical Arthroplasty for the Treatment of Cervical Degenerative Disc Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study progress and recruitment rate too low
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 05/25
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: Cervical; Disc; Arthroplasty; Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior Cervical Discectomy and Fusion (ACDF) (Other): Anterior Cervical Discectomy and Fusion with Cervical CFRP I/F CAGE® and SLIM LOC(R) Anterior Cervical Plate System with allograft
  Interventions: Device: ACDF
- Cervical Total Disc Replacement (Active Comparator): DISCOVER™ Artificial Cervical Disc
  Interventions: Device: DISCOVER™ Artificial Cervical Disc

INTERVENTIONS:
Device: DISCOVER™ Artificial Cervical Disc — DISCOVER™ Artificial Cervical Disc
  Arms: Cervical Total Disc Replacement
Device: ACDF — Cervical CFRP I/F CAGE® and SLIM LOC(R) Anterior Cervical Plate System with allograft
  Arms: Anterior Cervical Discectomy and Fusion (ACDF)

SUMMARY:
The purpose of the study is to evaluate the performance of the Discover cervical Artificial disc in the treatment of degenerative disc disease in one level of the cervical spine.

DETAILED DESCRIPTION:
The protocol underwent 3 amendments, the last of which (02APR2009) changed the study design from a randomized to a non-randomized and non-comparative clinical trial. All of the subjects were enrolled under the randomized design with the exception of the last subject. This study is not applicable per FDAA Title VIII, Section 801 due to the final trial design. However, results are submitted to clinicaltrials.gov due to the majority of study data being collected under a randomized (FDAA Title VIII, Section 801 applicable) trial design

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 18 and 65 years inclusive.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Objective evidence of cervical disc disease in one vertebral level between C3-C7 defined as one or more of the following:

  * Shoulder and/or arm pain in a radicular distribution resulting from herniated disc or bony osteophytes (Consistent w diagnostic imaging including Axial CT, CT Myelogram, MRI and/or plain films)
  * Subjects with myeloradiculopathy resulting from mild spinal cord compression and nerve root impingement
* Unresponsive to documented non-surgical management for ≥ 6 weeks and/or presents with progressive symptoms of nerve root or spinal cord compression in the face of continued non-surgical management (e.g., physical therapy, medication therapy, corticosteroid injections, etc.)
* Minimum Neck Disability Index score of ≥30 % (15/50 points)

Exclusion Criteria:

* Subjects who, in the opinion of the Clinical Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Subjects who are pregnant, lactating or wishes to become pregnant within the duration of the study.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical investigation with an investigational product in the last 30 days.
* Subjects who are currently involved in any injury litigation claims.
* Subjects with significant degeneration at more than one cervical level (e.g. DISH, ankylosing spondylitis, congenital abnormality, rheumatoid arthritis)
* Subjects who have had any prior surgery at the level to be treated (subjects with a prior Laminotomy at the level to be treated may be included in the study)
* Subjects who have marked cervical instability on lateral or flexion/extension x-rays defined as translation ≥3mm and/or ≥11 degrees of rotational difference to either adjacent level
* Subjects who have presence of systemic infection or infection at the site of surgery
* Subjects who have been diagnosed with malignancy
* Subjects who have been diagnosed with a condition or require postoperative medication(s) that may interfere with bony/soft tissue healing
* Subjects who have been diagnosed with Osteoporosis, Osteopenia, other metabolic bone disease or endocrine disorder known to affect osteogenesis.
* Subjects with pre-existing neurological abnormalities other than deficits produced from the spinal lesion (e.g., MS, Parkinson's, CVA, diabetic neuropathy, peripheral neuropathy).
* Subjects with morbid obesity defined as a BMI of ≥40, or more than 100 lbs (45.4kg) over ideal weight.
* Subjects with any known allergy to titanium metal, polyethylene, metal alloy or carbon fibre reinforced polymer
* Subjects who have had prior fusion surgery at any level(s) (C1-T1)
* Subjects with kyphosis >-15 degrees evaluated using the Cobb angle measurement
* Subjects with Significant cervical degenerative disease characterized by bridging anterior osteophytes, significant loss of disc space height (3mm or less), sclerotic facets, large posterior osteophytes, autofusion of other cervical levels, and degenerative retrolisthesis. Spinal diseases such as DISH, ankylosing spondylitis, congenital abnormality, and rheumatoid arthritis, should also be excluded
* Subjects undergoing treatment with a bone growth stimulator, which cannot be discontinued prior to enrollment in the study.
* Significant kyphotic deformity or significant reversal of lordosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - Westmead Private Hospital, Sydney, New South Wales
  - Calvary Hospital, Tasmania
- Klinikum Neustadt, Neustadt, Holstein, Germany
- Divisione di Neurochirurgia, Rome, Italy
- Island Hospital, George Town, Malaysia
- Elisabeth Ziekenhuis, Tilburg, Netherlands
- La Paz Hospital, Madrid, Spain
- Hope Hospital, Manchester, Lancashire, United Kingdom

REFERENCES:
- [Derived] Salmons HI, Galetta MS, Divi SN, Fried TB, Fang T, Hoffman E, Goyal DKC, Mangan JJ, Schroeder GD, Vaccaro AR. Are Industry-funded Studies of Cervical Disc Arthroplasty Versus Anterior Cervical Discectomy and Fusion Biased? Clin Spine Surg. 2021 Feb 1;34(1):1-3. doi: 10.1097/BSD.0000000000000946. No abstract available. PMID 32049677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 sites enrolled 60 subjects who were randomized into two treatment groups. Site 12 (17 subjects total) transferred into the Discover IDE study. Site 04 (5 subjects total) did not submit data, which was limited, due to EDC technical difficulties at the site. Therefore 38 subjects are reported in this study.
Groups:
- Cervical Total Disc Replacement: DISCOVER Artificial Cervical Disc
- ACDF: Anterior Cervical Discectomy and Fusion (ACDF)
Period: Overall Study
Arm/Group | Cervical Total Disc Replacement | ACDF
Started | 22 | 16
Completed | 18 | 12
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Total Disc Replacement | ACDF | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (8.87) | 47.5 (8.17) | 46.2 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  Spain | 2 | 1 | 3
  Germany | 0 | 1 | 1
  United Kingdom | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Success
Description: Overall success was a composite endpoint determined by the following clinical outcome measures: 1. Neck Disability Index ≥ 15-point improvement from baseline to 12 months post-operative, 2. No new clinically significant permanent abnormalities in neurological function (i.e. motor strength, nerve root tension signs, sensory and reflex signs) from baseline to 12 months post-operative, 3. No subsequent secondary surgical interventions (SSI) at the index level, and 4. No device-related serious events (dSAE) from intra-operative through 12-months post-operative. Please note that these time periods were intended to be from baseline to 24 months post-operative, but since the study was terminated early the 12 month time periods were utilized.
Time Frame: 12 months
Population: Overall Patient Success is composed of several outcome measures, some of which require a valid pre-operative and 12-month post-operative score. Due to withdrawals and incomplete or unavailable assessments, 18 subjects in the CTDR and 11 subjects in the ACDF treatment groups were available for the Overall Patient Success calculation.
Measure: Number; unit: Percentage of subjects
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
Percentage of subjects | 33.33 | 90.91

2. Secondary Outcome: Change in Visual Analogue Scale (VAS) Neck Pain From Pre-treatment to 12 Months
Description: The visual analogue scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 100 = 10 cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their neck.
Time Frame: 12 months
Population: Due to withdrawals and incomplete or unavailable assessments, 18 subjects in the CTDR and 11 subjects in the ACDF treatment groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
units on a scale | -16.6 (34.2) | -52.1 (22.86)

3. Secondary Outcome: Change in Visual Analogue Scale (VAS) Left Arm Pain From Pre-treatment to 12 Months.
Description: The visual analogue scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 100 = 10 cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their left arm.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
units on a scale | -15.9 (25.7) | -46.6 (43.5)

4. Secondary Outcome: Change in Visual Analogue Scale (VAS) Right Arm Pain From Pre-treatment to 12 Months.
Description: The visual analogue scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0= 0 cm) listed on the left and 'Very severe pain' (score of 100= 10 cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their right arm.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
units on a scale | -18.4 (32.8) | -20.5 (25.8)

5. Secondary Outcome: Change in Visual Analogue Scale (VAS) Right Shoulder Pain From Pre-treatment to 12 Months.
Description: The visual analogue scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 100 = 10 cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their right shoulder.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
units on a scale | -15.7 (35.4) | -22.4 (32.7)

6. Secondary Outcome: Change in Visual Analogue Scale (VAS) Left Shoulder Pain From Pre-treatment to 12 Months.
Description: The visual analogue scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 10 = 10 cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their left shoulder.
Time Frame: 12 Months
Population: Due to withdrawals and incomplete or unavailable assessments, 17 subjects in the CTDR and 11 subjects in the ACDF treatment groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 17 | 11
units on a scale | -17.1 (28.9) | -49.8 (36.5)

7. Secondary Outcome: Change in Mental Component Summary Quality of Life Measure Assessed by Short Form SF-36 From Pre-treatment to 12 Months
Description: The 36-item Short Form Health Survey (SF-36) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-36) and Mental Component Score (MCS-36)
Time Frame: 12 months
Population: Due to withdrawals and incomplete or unavailable assessments, 16 subjects in the CTDR and 10 subjects in the ACDF treatment groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 16 | 10
units on a scale | 4.1 (13.2) | 15.1 (14)

8. Secondary Outcome: Change in Physical Component Summary Quality of Life Measure Assessed by Short Form SF-36 From Pre-treatment to 12 Months
Description: as for outcome 7
Time Frame: 12 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 16 | 10
units on a scale | 8.1 (11.7) | 17.7 (9.2)

9. Secondary Outcome: Change in Function Assessed by Neck Disability Index Improvement From Pre-treatment to 12 Months
Description: The neck disability index (NDI) is a validated, disease specific, self-administrated questionnaire for assessing pain intensity and function in patients with neck pain on a scale from 0 to 100. A lower score is a better result (i.e. less severe pain and/or better function). The proportion of patients with an improved score (lower) of 15 points or more was the analysis variable.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Subjects
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 11
Percentage of Subjects | 33.33 | 90.91

10. Secondary Outcome: Work Status Assessed at 12 Months
Description: The proportion of subjects with unrestricted work status (compared to subjects not working or with restricted work status) is reported at the 12 month follow-up interval.
Time Frame: 12 months
Population: Due to withdrawals and incomplete or unavailable assessments, 18 subjects in the CTDR and 12 subjects in the ACDF treatment groups were available for this outcome.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 18 | 12
Percentage of Subjects | 38.89 | 50.00

11. Secondary Outcome: Sagittal Angulation, Also Known as Global Lordosis, Measured Radiographically at 6 Months
Description: Sagittal Angulation is a measure of the angle formed between the inferior endplate of the C2 vertebrae and the corresponding inferior endplate of vertebrae C7 of the spine, measured in degrees, from a side (sagittal) view.
Time Frame: 6 months
Population: Only 2 subjects in the Cervical Total Disc Replacement (cTDR) and 1 subject in the ACDF treatment groups were available for this outcome measure. There were 2 ACDF subjects at this endpoint, however one subject was missing the flexion extension rotation radiographic view therefore could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 2 | 1
degrees | 9.6 (10) | -1.5 (NA) — One ACDF subject was missing the flexion extension rotation radiographic view therefore could not be included in the analysis.

12. Secondary Outcome: Adjacent Level Degeneration Measured Radiographically at 24 Months
Description: Adjacent Level Degeneration is evaluated using a point system that assigns numerical scores to severity of Height Loss, Anterior Osteophytes, and Endplate Sclerosis; and then grades into one of the following five categories: None, Mild, Moderate, Severe, or NA.
Time Frame: 24 months
Population: Study was terminated prior to 24 months therefore there are no results for this endpoint.
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Maintenance of Disc Height Measured Radiographically at 6 Months
Description: Maintenance of disc height is measured at the index and adjacent levels to determine the effect of the treatment on restoration or maintenance of the disc height. Initial post-operative disc height is compared with subsequent post-operative visits (i.e. 6 months) to evaluate the maintenance of disc height. The height is measured in millimeters (mm).
Time Frame: 6 months
Population: Only 2 subjects in the cTDR and 1 subject in the ACDF treatment groups were available for this outcome measure. There were 2 ACDF subjects at this endpoint, however one subject was missing the flexion extension rotation radiographic view therefore could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 2 | 1
mm | 4.7 (0.57) | 5.1 (NA) — One ACDF subject was missing the flexion extension rotation radiographic view therefore could not be included in the analysis

14. Secondary Outcome: Foraminal Height Measured Radiographically at 24 Months
Description: Foraminal height is the maximum vertical distance, measured in millimeters (mm), between the inferior surface of the superior pedicle and superior surface of the inferior pedicle. These measurements are obtained via magnetic resonance imaging (MRI).
Time Frame: 24 months
Population: The study was terminated prior to 24 months therefore there are no results for this endpoint.
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Cervical Range of Motion Measured Radiographically at 6 Months
Description: Cervical range of motion measures the angle, in degrees, between the inferior endplate of C2 to the inferior endplate of C7 on flexion-extension radiographs.
Time Frame: 6 months
Population: Only 2 subjects in the cTDR and 2 subjects in the ACDF treatment groups were available for this outcome measure.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 2 | 2
degrees | 53.9 (16.4) | 55.2 (25.5)

16. Secondary Outcome: Device Related Adverse Events
Description: The proportion of subjects with device related adverse events as reported throughout the duration of the study.
Time Frame: Intra-operatively to 24 months post-operative
Measure: Number; unit: Percentage of subjects
Arm/Group | Cervical Total Disc Replacement | ACDF
Number analyzed (Participants) | 22 | 16
Percentage of subjects | 13.64 | 0.00

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the intra-operatively to 24 months post-operative timepoint (the patient with the longest follow-up for potential AE reporting was 24 months).
Arm/Group | Cervical Total Disc Replacement | ACDF
Serious Adverse Events (participants affected / at risk) | 3/22 | 1/16
Other Adverse Events (participants affected / at risk) | 9/22 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Total Disc Replacement (N=22) | ACDF (N=16)
Lower Respiratory Tract Infections (Infections and infestations) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Total Disc Replacement (N=22) | ACDF (N=16)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Horner's Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early therefore the latest clinical data available is at the 12 month post-operative timepoint and the latest radiographic data available is at the 6 month post-operative timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after DePuy has been given the opportunity of reviewing the proposed presentation or publication at least 30 days prior to the intended submission, presentation, or publication date.